CLINICAL TRIAL: NCT02383030
Title: Randomized Phase III Study of Fulvestrant as Maintenance Therapy After First-line Chemotherapy in HER2 Negative Postmenopausal Metastatic Breast Cancer Patients
Brief Title: Fulvestrant as Maintenance Therapy After First-line Chemotherapy in HER2 - Postmenopausal MBC Patients
Acronym: FUMANCE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Consorzio Oncotech (Other)
Collaborators: Clinical Research Technology S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: GIM18-FUMANCE; 2014-003798-41 (EudraCT Number)
Record Dates: First submitted 2015-02-26; First posted 2015-03-09 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-06

CONDITIONS: Metastatic Breast Cancer
Keywords: Breast cancer; Metastatic; HER2 negative; postmenopausal; maintenance therapy; fulvestrant
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fulvestrant (Experimental): In Arm A maintenance Fulvestrant will be given until disease progression, unacceptable toxicity or refused of patient to the treatment.
  Interventions: Drug: Fulvestrant
- No intervention (No Intervention): Patients will be randomized to receive fulvestrant (experimental arm) or no treatment

INTERVENTIONS:
Drug: Fulvestrant — After randomization patients will receive (Arm A, experimental Arm) fulvestrant as the following schedule: 500 mg i.m. on Days 0, 14, 28 followed by fulvestrant 500 mg im given every 28 days until progression disease. Study will start after 42 days from the last cycle of chemotherapy
  Other Names: Faslodex
  Arms: Fulvestrant

SUMMARY:
Breast cancer is one of the most prevalent cancers among women, and represents 20 - 25% of all female cancers. Despite earlier diagnosis and improvement in adjuvant therapies, some patients will present metastatic recurrence.

Treatment of breast cancer is determined by the extent of the disease. Early or localized breast cancer is treated by a combination of surgery and radiotherapy. Adjuvant systemic therapy, consisting of chemotherapy and/or endocrine therapy, in tumors deemed hormone responsive, can prolong the disease-free interval and improve overall survival. However, approximately 30% to 40% of patients with early breast cancer will ultimately relapse, with either local recurrence or distant metastases, and require further systemic treatment for advanced disease.

Since breast cancer that recurs or progresses after initial treatment is considered incurable, the therapy options available for advanced disease are concerned with disease control and palliation of symptoms.

Hormonal therapy has become the treatment of choice in postmenopausal women with hormone sensitive breast cancer. Even though the treatment of advanced breast cancer in postmenopausal women has improved with the introduction of agents such as aromatase inhibitors, these agents still have limitations, and disease management continues to be sub-optimal. The use of systemic therapies such as hormonal therapy, chemotherapy or new biological treatment is to reduce tumour masses, improve survival and preserve quality of life. Whatever the initial efficacy of the treatment undertaken in metastatic setting, almost every patient will relapse. The main goal is to improve progression free survival (PFS). To achieve this, the type of chemotherapy, the optimal duration of chemotherapy, the benefit of maintenance chemotherapy, the benefit of maintenance hormonal treatment are debatable.

DETAILED DESCRIPTION:
The search for prognostic and predictive factors that could influence the survival of patients treated for metastatic breast cancer has already been the subject of several studies. It seems that 2 components in the natural outcome of tumors must be considered. The first category is related to the primary characteristics such as initial histological grade, hormonal receptor status. The second category is linked to the metastatic characteristics: proliferation index reflected by the length of disease-free interval, type and number of metastatic sites involved. On the other hand, some prognostic factors are linked to the treatments undertaken, stressing their impact on the natural outcome of the disease: type of hormonotherapy, type of chemotherapy, type of response achieved by treatment.

The impact of some factors remains debatable, such the duration of treatment. The optimal duration of chemotherapy in patients who respond or have stable disease is not identified.

Definitively, the major limit to the use of prolonged regimens of chemotherapy is related to their toxicity, all the more so as they are cumulative (cardiac toxicity of anthracyclins, neurologic toxicity of taxanes, haematological cumulative toxicities with any chemotherapy…). The proposition to give hormonal treatment to prolong therapy in hormonal-positive tumors is another possible option. In the literature, data focused on this strategy are rare.

One can object that the choice of patient/tumor characteristics for who would or would not receive the maintenance hormonal therapy was not random, or controlled in any way. This may have led to a selection of better prognosis patients. Investigators cannot know whether they are observing natural history or impacting it in such a trial. Nevertheless the major impact obtained by maintenance hormonal treatment after the first line chemotherapy might indicate that this strategy should be recommended in patients with an ER or PgR positive tumor. Based on the amplitude of the benefit observed, it may be ethically debatable to conduct a prospective randomized study. Moreover, randomized trials which assess the benefit of a new chemotherapy regimen should allow the possibility to give maintenance hormonal treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically diagnosis of breast cancer;
2. Presence of metastatic disease either measureable or non-measureable but evaluable bone disease as defined by the Response Evaluation Criteria in Solid Tumors;
3. Diagnosis of hormone receptor positive (HR+), HER2 negative breast cancer. To fulfill the requirement for HR+ disease, a breast cancer must express, by immunohistochemistry (IHC), at least one of the hormone receptors (estrogen receptor [ER], progesterone receptor [PR]). To fulfill the requirement for HER2 negative disease, a breast cancer must not demonstrate over-expression of HER2 by either IHC or fluorescence in-situ hybridization (FISH);
4. Post-menopausal status at the time of randomization.
5. Previous treatment with either an antiestrogen or an aromatase inhibitor for adjuvant or metastatic disease is allowed;
6. Age >18;
7. One line chemotherapy for metastatic disease discontinued for 21-28 days. Patient has to have response or stability from the first-line chemotherapy. The patient may have received prior systemic chemotherapy in the neo-adjuvant or adjuvant setting;
8. Patients with measurable or evaluable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria;
9. Performance Status (ECOG) <2;
10. No brain metastases;
11. No clinically serious concurrent illnesses;
12. Adequate organ function
13. Use of bisphosphonates are allowed;
14. Use of antiangiogenetic drugs (bevacizumab associated to paclitaxel) is allowed, but discontinued 21-28 days before start study;
15. Life expectancy > 12 weeks;
16. Are willing to participate for the duration of the study and to follow study procedures;
17. Written informed consent prior to any study-specific procedures Written informed consent;

Exclusion Criteria:

1. Treatment with a drug that has not received regulatory approval for any indication within 21-28 days from the randomization;
2. Drug (chemotherapy or biological drug) after the end of first-line chemotherapy for maintenance phase;
3. Significant known cardiovascular impairment (NYHA CHF > grade 2, unstable angina, myocardial infarction within the previous 6 months prior to randomization, or existing serious cardiac arrhythmia). VECF (Ventricular Ejection Cardiac Fraction) ≤ 50%;
4. Prior malignancy (other than breast cancer) except for non-melanoma skin cancer and carcinoma in situ (of the cervix or bladder), unless diagnosed and definitively treated more than 5 years prior to randomization;
5. Severe/uncontrolled intercurrent illness within the previous 28 days prior to randomization.
6. Any other significant co-morbid conditions that in the opinion of the Investigator would impair study participation or cooperation;
7. Patients with psychiatric illness, social situation or geographical situation that would preclude informed consent or limit compliance with study requirements, as determined by the Investigator;

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-09 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Maintenance-progression-free survival (mPFS) | 36 months
  Time between the date of randomization and the date of progression or death, whichever occurs first

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Cognetti, Study Chair — Regina Elena National Cancer Institute Via Elio Chianesi 53, 00144 Rome, Italy
Locations (20):
- Italy (20):
  - A.S.U.R. Zona Territoriale 6 Fabriano U.O. Oncologia Medica, Fabriano, Ancona
  - A.S.L. LT - Ospedale Santa Maria Goretti U.O.C. di Oncologia Medica, Latina, Latina
  - Ospedale Unico Versilia U.O. Oncologia Medica, Lido di Camaiore, Lucca
  - Presidio Ospedaliero di Macerata, Mecerata, MC
  - Istituto Nazionale dei Tumori - Fondazione G. Pascale U.O. Oncologia Medica Senologica, Napoli, Napoli
  - Ospedale 'Felice Lotti' - Azienda USL 5 di Pisa U.O. di Oncologia Medica, Pontedera, Pisa
  - Ospedale Oncologico Regionale - Centro di Riferimento Oncologico di Basilicata U.O. di Oncologia Medica, Rionero in Vulture, Potenza
  - Istituto Regina Elena per lo studio e la cura dei tumori S.C. Oncologia Medica A, Roma, Roma
  - Ospedale C. e G. Mazzoni di Ascoli Piceno - Area Vasta 5, Ascoli Piceno
  - P.O. Avezzano Via G. di Vittorio, 6, Avezzano
  - Ospedale degli Infermi - Faenza, Faenza
  - A.O.U Ospedali Riuniti di Foggia, Foggia
  - Ospedale Vito Fazzi, Lecce
  - P.O. Campo di Marte, Lucca
  - Azienda Ospedaliera Fatebenefratelli e Oftalmico, Milan
  - Università di Napoli Federico II Dipartimento di Medicina clinica e Chirurgia, Naples
  - A.O.R.N. "A. Cardarelli", Napoli
  - Ospedale di Ravenna, Ravenna
  - Ospedale fatebenefratelli - Villa S Pietro (Roma), Roma
  - Ospedale civile "Madonna del Soccorso" - Area Vasta 5, San Benedetto del Tronto

IPD SHARING:
Plan to Share IPD: No